CLINICAL TRIAL: NCT04971057
Title: The Effects of Multimedia Information for Patients With Renal Biopsy
Brief Title: Multimedia Information for Patients With Renal Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ching-Hui Chien, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201900682B0C
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Pain; Anxiety; Hematuria
Keywords: multimedia information; renal biopsy; self-efficacy; pain; anxiety; positive and negative affective; hematuria
MeSH Terms: conditions — Pain; Anxiety Disorders; Hematuria

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group received routine care
- Multimedia information Group (Experimental): The experimental group received a multimedia information
  Interventions: Other: multimedia information program of renal biopsy

INTERVENTIONS:
Other: multimedia information program of renal biopsy — Multimedia information program is based on self-efficacy theory. The multimedia videos contain the information associated with renal biopsy, which including the purpose, indications, preparations for the examination, process, patient experience sharing, complications, precautions, home care and stress adjustment strategies.
  Arms: Multimedia information Group

SUMMARY:
This study takes place in the Divisions of Nephrology. Patients undergoing renal biopsy were randomized to control group or multimedia information intervention group. The control group received routine care, and the multimedia information intervention group received a multimedia information. After the pre-test, the two groups performed the 1 to 3 post-tests on pre-operation, post-operative day 1 and post-operative day 9. This study used questionnaires that including General Self-Efficacy Scale, Pain Visual Analogy Scale, Visual Analogue Scale for Anxiety, and Positive and Negative Affective Scale.

DETAILED DESCRIPTION:
This study takes place in the Divisions of Nephrology at Chang Gung Memorial Hospitals. Patients undergoing renal biopsy were randomized to control group or multimedia information intervention group. The control group received routine care, and the multimedia information intervention group received a multimedia information. Multimedia information intervention is based on self-efficacy theory. The multimedia videos contain the information associated with renal biopsy, which including the purpose, indications, preparations for the examination, process, patient experience sharing, complications, precautions, home care and stress adjustment strategies. In addition, the investigator also provide face-to-face consultations on answers and clarifications for the content of the videos and telephone consultations to understand the self-care situation of patients on the third day after discharge. After the pre-test, the two groups performed the 1 to 3 post-tests on pre-operation, post-operative day 1 and post-operative day 9. This study used questionnaires that including General Self-Efficacy Scale, Pain Visual Analogy Scale, Visual Analogue Scale for Anxiety, and Positive and Negative Affective Scale. Generalized Estimating Equations (GEEs) will be used to o analyze data.

ELIGIBILITY:
Inclusion Criteria:

1. patients are at least 20 years old
2. patients need to undergo a renal biopsy
3. patients can communicate in Chinese or Taiwanese
4. patients agree to participate in the research and sign the consent form
5. patients have family members accompanying

Exclusion Criteria:

1. patients have undergone renal biopsy before
2. patients have history of mental disorder
3. patients use anticoagulants

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-14 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
General Self-Efficacy Scale | pretest
  A total of 10 items. A 4-point(1-4) scoring method was adopted. Higher scores indicate higher self-efficacy
General Self-Efficacy Scale | post-operative day 9
  A total of 10 items. A 4-point(1-4) scoring method was adopted. Higher scores indicate higher self-efficacy
Pain Visual Analogy Scale | pretest
  It is an actual straight line of 100 mm, of which 0 mm means no pain at all and 100 mm means extreme pain. A higher score indicates greater pain intensity
Pain Visual Analogy Scale | pre-operation
  It is an actual straight line of 100 mm, of which 0 mm means no pain at all and 100 mm means extreme pain. A higher score indicates greater pain intensity.
Pain Visual Analogy Scale | post-operative day 1
  It is an actual straight line of 100 mm, of which 0 mm means no pain at all and 100 mm means extreme pain. A higher score indicates greater pain intensity.
Pain Visual Analogy Scale | post-operative day 9
  It is an actual straight line of 100 mm, of which 0 mm means no pain at all and 100 mm means extreme pain. A higher score indicates greater pain intensity.
Visual Analogue Scale for Anxiety | pretest
  It is an actual straight line of 100 mm, of which 0 mm means no anxiety at all and 100 mm means extreme anxiety. A higher score indicates greater severity of anxiety
Visual Analogue Scale for Anxiety | pre-operation
  It is an actual straight line of 100 mm, of which 0 mm means no anxiety at all and 100 mm means extreme anxiety. A higher score indicates greater severity of anxiety
Visual Analogue Scale for Anxiety | post-operative day 1
  It is an actual straight line of 100 mm, of which 0 mm means no anxiety at all and 100 mm means extreme anxiety. A higher score indicates greater severity of anxiety
Visual Analogue Scale for Anxiety | post-operative day 9
  It is an actual straight line of 100 mm, of which 0 mm means no anxiety at all and 100 mm means extreme anxiety. A higher score indicates greater severity of anxiety

SECONDARY OUTCOMES:
Positive and Negative Affective Scale | pretest
  It contains a total of 20 items with two subscales including positive affective subscale and negative affective subscale. A 4-point (1-4) scoring method is used. Higher scores represent higher levels of positive and negative affect
Positive and Negative Affective Scale | post-operative day 9
  It contains a total of 20 items with two subscales including positive affective subscale and negative affective subscale. A 4-point (1-4) scoring method is used. Higher scores represent higher levels of positive and negative affect

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital at Linkou, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akca A, Yilmaz G, Esmer AC, Yuksel S, Koroglu N, Cetin BA. Use of video-based multimedia information to reduce anxiety before office hysteroscopy. Wideochir Inne Tech Maloinwazyjne. 2020 Jun;15(2):329-336. doi: 10.5114/wiitm.2019.89378. Epub 2019 Oct 28. PMID 32489494
- [Background] Batuyong ED, Jowett AJ, Wickramasinghe N, Beischer AD. Using multimedia to enhance the consent process for bunion correction surgery. ANZ J Surg. 2014 Apr;84(4):249-54. doi: 10.1111/ans.12534. PMID 24812709
- [Background] Bowers N, Eisenberg E, Montbriand J, Jaskolka J, Roche-Nagle G. Using a multimedia presentation to improve patient understanding and satisfaction with informed consent for minimally invasive vascular procedures. Surgeon. 2017 Feb;15(1):7-11. doi: 10.1016/j.surge.2015.09.001. Epub 2015 Oct 14. PMID 26464072
- [Background] Brachemi S, Bollee G. Renal biopsy practice: What is the gold standard? World J Nephrol. 2014 Nov 6;3(4):287-94. doi: 10.5527/wjn.v3.i4.287. PMID 25374824
- [Background] Chung S, Koh ES, Kim SJ, Yoon HE, Park CW, Chang YS, Shin SJ. Safety and tissue yield for percutaneous native kidney biopsy according to practitioner and ultrasound technique. BMC Nephrol. 2014 Jun 23;15:96. doi: 10.1186/1471-2369-15-96. PMID 24957046
- [Background] Demircelik MB, Cakmak M, Nazli Y, Sentepe E, Yigit D, Keklik M, Arslan M, Cetin M, Eryonucu B. Effects of multimedia nursing education on disease-related depression and anxiety in patients staying in a coronary intensive care unit. Appl Nurs Res. 2016 Feb;29:5-8. doi: 10.1016/j.apnr.2015.03.014. Epub 2015 Apr 7. PMID 26856480
- [Background] D'Souza V, Blouin E, Zeitouni A, Muller K, Allison PJ. Multimedia information intervention and its benefits in partners of the head and neck cancer patients. Eur J Cancer Care (Engl). 2017 Jul;26(4). doi: 10.1111/ecc.12440. Epub 2016 Jan 18. PMID 26777257
- [Background] Ellett L, Villegas R, Beischer A, Ong N, Maher P. Use of a multimedia module to aid the informed consent process in patients undergoing gynecologic laparoscopy for pelvic pain: randomized controlled trial. J Minim Invasive Gynecol. 2014 Jul-Aug;21(4):602-11. doi: 10.1016/j.jmig.2014.01.002. Epub 2014 Jan 23. PMID 24462856
- [Background] El-Reshaid K, El-Reshaid W, Al-Bader D, Varro J, Madda J, Sallam HT. Biopsy of small kidneys: A safe and a useful guide to potentially treatable kidney disease. Saudi J Kidney Dis Transpl. 2017 Mar-Apr;28(2):298-306. doi: 10.4103/1319-2442.202767. PMID 28352011
- [Background] Hirsch JK, Sirois FM, Molnar D, Chang EC. Pain and Depressive Symptoms in Primary Care: Moderating Role of Positive and Negative Affect. Clin J Pain. 2016 Jul;32(7):562-7. doi: 10.1097/AJP.0000000000000292. PMID 26379073
- [Background] Hsueh FC, Chen CM, Sun CA, Chou YC, Hsiao SM, Yang T. A Study on the Effects of a Health Education Intervention on Anxiety and Pain During Colonoscopy Procedures. J Nurs Res. 2016 Jun;24(2):181-9. doi: 10.1097/jnr.0000000000000112. PMID 26551213
- [Background] Hu T, Liu Q, Xu Q, Liu H, Feng Y, Qiu W, Huang F, Lv Y. Absorption fever characteristics due to percutaneous renal biopsy-related hematoma. Medicine (Baltimore). 2016 Sep;95(37):e4754. doi: 10.1097/MD.0000000000004754. PMID 27631225
- [Background] Karadag E. The effect of a self-management program on hand-washing/mask-wearing behaviours and self-efficacy level in peritoneal dialysis patients: a pilot study. J Ren Care. 2019 Jun;45(2):93-101. doi: 10.1111/jorc.12270. Epub 2019 Mar 2. PMID 30825408
- [Background] Kauric-Klein Z, Peters RM, Yarandi HN. Self-Efficacy and Blood Pressure Self-Care Behaviors in Patients on Chronic Hemodialysis. West J Nurs Res. 2017 Jul;39(7):886-905. doi: 10.1177/0193945916661322. Epub 2016 Jul 24. PMID 27456461
- [Background] Mohammed A, Manjanabil P, deTakats D. Retroperitoneum: a forgotten and fatal aspect of kidney biopsy. Saudi J Kidney Dis Transpl. 2014 Nov;25(6):1278-81. doi: 10.4103/1319-2442.144267. PMID 25394450